CLINICAL TRIAL: NCT02409082
Title: The Presence of Pre-Alzheimers/Alzheimers Disease (AD) and Neuromarkers Related to Morbidity/Mortality in Patients With Acute Hip Fractures
Brief Title: Alzheimers Disease and Neuromarkers in Patients With Acute Hip Fractures
Acronym: ADhipfract
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Associate professor/MD/PhD, Sahlgrenska University Hospital
Other Study IDs: HOFTDEM
Record Dates: First submitted 2015-03-25; First posted 2015-04-06 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Alzheimers Disease; Inflammation; Hip Fracture
MeSH Terms: conditions — Alzheimer Disease; Inflammation; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — AD correlated factors like betamayloid and tau as well as interleukins
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators explore the presence of AD factors beta-amyloid and tau in CSF and plasma to verify AD diagnosis in patients with acute hip fracture. Clinical dementia test is performed prior to operation. Blood samples and CSF samples are collected at surgery and blood samples are collected postoperatively at intervals. Mortality is assessed at 30 days, 3 months and 1 year. Morbidity is assessed at , 3 months and >1 year. Neuromarkers specifically addressing the inflammatory component are to be analyzed and correlated to outcome together with AD markers, as above.

DETAILED DESCRIPTION:
The hypotheses explored in this investigation is that patients being pre-AD or having AD have worse prognosis following an acute hip fracture. This has been demonstrated in retrospective studies. In this study we admit all patients with a hip fracture planned tro receive a spinal anesthesia. Our golden standard of anesthesia in this patient cohort. Preoperatively Clinical Dementia Score is assessed after study inclosure. At the performance of the spinal dosage is standardized. Prior to giving this 5 ml of CSF is collected and blood is collected. Blood is then collected at intervals up until day 3 postoperatively. We plan to analyze beta-amyloid and tau in CSF and plasma to verify AD diagnosis in patients with acute hip fracture. Mortality is assessed at 30 days, 3 months and 1 year. Morbidity is assessed at, 3 months and >1 year. Neuromarkers specifically addressing the inflammatory component are to be analyzed and correlated to outcome together with AD markers, as above.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture with a planed spinal anesthesia

Exclusion Criteria:

* Not receiving a spinal anesthesia i.e. no CSF is available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with an acute hip fracture receiving a spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Mortality and morbidity | 1year
  interview by phone and death registration

CONTACTS AND LOCATIONS:
Overall Officials: Bengt M Nellgard, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Västra Götaland County, Sweden